CLINICAL TRIAL: NCT02522533
Title: Intervention for Pre-Frailty and Frailty in Thoracic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0192
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Therapy (Experimental): Patients will be receiving 6 weeks of an exercise program.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — 6 weeks of an exercise program.

SUMMARY:
Frailty has been associated with poor acute and long-term outcomes after major surgery. We recently determined that nearly 70% of patients undergoing major thoracic surgery are pre-frail or frail. We are interested in assessing whether a strength training intervention for frail or pre-frail patients has an impact on surgical decision making and on surgical outcomes.

ELIGIBILITY:
Inclusion Criteria: • Age ≥60 years, • Qualified to consent for participation in a research study, •Thoracic disease that may require major surgery (major anatomic lung resection, esophagectomy, repair of giant paraesophageal hernia, chest wall resection, extended pleurectomy/decortication, thymectomy or major surgery for other mediastinal process),• No obvious contraindications to surgery (end-stage heart disease, end-stage lung disease, severe dementia, other specific comorbidity that would prevent surgery), • Ability to participate in physical therapy and an independent exercise program for frailty mitigation, •No need for induction chemotherapy or radiation therapy, • Recent evaluation including computed tomography of the chest or chest/abdomen.

Exclusion Criteria:• Age <60 years, •Unable to provide informed consent, • No indication for major thoracic surgery, •Obvious contraindication to major thoracic surgery (end-stage heart disease, end-stage lung disease, severe dementia, other specific comorbidity that would preclude surgery),• Inability to participate in physical therapy and/or an independent home exercise for frailty mitigation, •Need for induction chemotherapy or radiation therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Reduction in the degree of frailty after strength training | 18 months

SECONDARY OUTCOMES:
Changes in surgeon risk assessment after strength training | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ferguson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States